CLINICAL TRIAL: NCT06334354
Title: Cognitive Aging in Older Long-term Breast Cancer Survivors
Brief Title: A Study of Changes in Thinking Related to Aging and Cancer in Breast Cancer Survivors (TRAC)
Acronym: TRAC
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-320
Record Dates: First submitted 2024-03-19; First posted 2024-03-28 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Survivors
Keywords: Cognitive aging
MeSH Terms: interventions — Restraint, Physical; Apolipoproteins E

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salvia, Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Survivor (BCS): Enrolled participants will be asked to complete a one-time, remote neurocognitive assessment. The neurocognitive assessment will consist of the CogSuite Neurocognitive Battery, an online, remotely deliverable battery of cognitive experimental measures, and a standard battery of remote neuropsychological measures. DNA will be collected via mailed saliva kits to assess Apolipoprotein E (APOE) status.
  Interventions: Other: Assessments; Other: Assessment (Survivors Only); Other: APOE and DNA Isolation
- Non-cancer Control (NCC): Enrolled participants will be asked to complete a one-time, remote neurocognitive assessment. The neurocognitive assessment will consist of the CogSuite Neurocognitive Battery, an online, remotely deliverable battery of cognitive experimental measures, and a standard battery of remote neuropsychological measures. DNA will be collected via mailed saliva kits to assess Apolipoprotein E (APOE) status.
  Interventions: Other: Assessments; Other: APOE and DNA Isolation

INTERVENTIONS:
Other: Assessments — Sociodemographics, Deficit Accumulation Questionnaires, Remote Cognitive Assessment, Deficit Accumulation Questionnaires,Remote Cognitive Assessment
Other: Assessment (Survivors Only) — *Tumor/Treatment Variables (Survivors Only)
  Groups: Breast Cancer Survivor (BCS)
Other: APOE and DNA Isolation — Biospecimens procurement and processing

SUMMARY:
The purpose of this study is to look at how differences in cognitive (mental) function develop over time in breast cancer survivors compared to volunteers without a history of cancer (healthy volunteers). Both cancer survivors and healthy volunteers (who are the same age as the cancer survivors) will participate in this study so the researchers can compare the results of neurocognitive testing (which looks at memory, attention, and information processing) on each group of participants.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Per medical record and/or self-report, identifies as female
* Per medical record and/or self-report, currently age 60-80
* Per self-report, has access to a computer and internet connectivity
* Score of <11 on Blessed Orientation-Memory-Concentration Test (BOMC)
* As per medical record or self-report, if currently taking psychoactive medications (including but not limited to antidepressants and anxiolytics), dose must have been stable at least two months prior to enrollment.
* English fluent (as per self-report, fluency of "well" or "very well", and having a reasonable comprehension of the study conversation in the opinion of the research staff)**

Breast Cancer Survivors:

* Per medical record and/or self-report, history of stage 0-3 breast cancer diagnosed between 50-60 years of age
* Per medical record and/or self-report, no evidence of disease (NED)

Non-Cancer Controls:

* Per self-report, no history of breast cancer

  * Language verification: For both survivors and controls, prior to enrollment, all will be asked the following two questions by a CRC to verify English fluency necessary for participation in the study:

    1. How well do you speak English? (must respond "Well" or "Very well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
    2. What is your preferred language for healthcare? (must respond English)

Exclusion Criteria:

All participants:

* As per medical record or self-report, diagnosis of neurodegenerative disorder that affects cognitive function (e.g. Alzheimer's disease, Parkinson's disease, Multiple Sclerosis, Dementia, Seizure Disorders, etc.)
* As per medical record or self-report, history of stroke or head injury resulting in a structural lesion on neuropsych imaging, persistent cognitive difficulties impacting work or daily life, or required cognitive rehabilitation
* As per medical record or self-report, a diagnosis of a major Axis I psychiatric disorder including Schizophrenia Spectrum Disorder, substance use disorder, Bipolar Disorder or Schizotypal personality disorder. Schizophrenia Spectrum Disorders include Schizophrenia, Schizophreniform disorder, Schizoaffective disorder, Delusional disorder, Brief psychotic disorder, and Attenuated Psychotic Disorder.
* As per medical record or self-report, visual or auditory impairment that would preclude ability to complete the assessments (e.g. history of significant macular degeneration or being unable to correct hearing with hearing aids)
* As per medical record or self-report, use of methotrexate (Amethopterin, Rhematrex, Trexall) or rituximab (Rituxin) for rheumatoid arthritis, psoriasis or Crohn's disease, or cyclophosphamide (Cytoxan, Neosar) for lupus.
* As per medical record or self-report, participation in a conflicting (overlapping neurocognitive assessments) research study (i.e. MSK 18-294)

Breast Cancer Survivors:

* As per medical record or self-report, history of cancer recurrence
* As per medical record or self-report, any history of another cancer except nonmelanoma skin cancer or first breast cancer (a secondary breast cancer is exclusionary)
* As per medical record or self-report, breast cancer only treated with surgery

Non-Cancer Controls:

* As per medical record or self-report, history of treatment using radiation, chemotherapy, and/or Tamoxifen or Aromatase-inhibitors
* As per medical record or self-report, any history of cancer except non-melanoma skin cancer

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Study Population: Survivors will be recruited in Breast Medicine Service clinics at the Breast and Imaging Center (BAIC) after having been identified via a Dataline query and/or weekly clinic schedules or through direct referrals from a member of the patient's treatment team.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
examine cognitive effects | within 45 days of participant consent
  of remote cancer diagnosis and treatment and potential association with increased/accelerated deficit accumulation in older survivors.The primary outcome is cognitive performance, as measured by CogSuite aggregate intra-individual variability, the average intra-individual variability across the subtests. Cognition will be assessed using the CogSuite battery of five subtests: 1) Attention Network Test; 2) Mental Rotation; 3) Stop Signal Delay; 4) N-back; and 5) Psychomotor Speed measures.

SECONDARY OUTCOMES:
measure levels of smoking exposure | within 45 days of participant consent
  by testing cotinine (an important metabolite of nicotine) in urine samples to examine possible interactions of smoking history with genetic variants, e.g., APOE ε4+, on cognition

CONTACTS AND LOCATIONS:
Overall Officials: James Root, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm